CLINICAL TRIAL: NCT06634329
Title: Assessment of the Comfort of Preterm Newborns During Feeding, Comparison of Different Methods of Milk Administration With Gastric Tube
Brief Title: Preterm Newborn's Behavioral Responses During Feeding With Gastric Tube
Acronym: PREMALIM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: CE-2024-56
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Premature Birth
Keywords: Preterm infants; Oro/nasogastric tube feeding; Developmental care; Parents integration
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oro or Nasogastric tube feeding — Parental involvement in their premature baby's feeding

SUMMARY:
Preterm infants need aims of a tube named oral or naso gastric to grow until they acquire autonomy in suction-swallowing.

In fact, several modes feed by a gastric tube exist : using an electric syringe pump (continuous administration), or manual and individualization administration. In this second case, milk can be delivered by gravity, depending on the height the syringe is placed above the infant, or by manually pushing on the syringe. Milk can be administrated by nurses or by the parents after a learning period.

In this observational study, we would like to compare the preterm infants' behavioral during these different naso or oro gastric feeding modes by observing well-being signs and withdrawal signs (Dsilna grid) on video settings.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at the University Hospitals of Strasbourg during October 2024 and October 2025
* Needing nasogastric tube feeding during at least 4 days
* With parents (legal representants) having expressed their agreement with the use of video recording in the framework of the current study

Exclusion Criteria:

* ORL malformations
* Neurological dysfunction
* Sedated infant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborn infants needing nasogastric tube feeding hospitalized at Rénaimation et médecine du nouveau né / University Hospital of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Comparing the tolerance of these different types of food (gravity versus pushing the seringue), based on the child's behavioral and physiological signs of well-being. | 6 months
  Observation of preterm infants during and after naso/oro gastric tube feeding on videos to record well-being and withdrawal signs like classified in the Dsilna grid every 4 minutes.

SECONDARY OUTCOMES:
- Well-being and withdrawal signs by the Dsilna grid : comparison of manual methods versus electric syringe administration | 6 monts
  Comparaison of the score of withdrawal or well being tube in this different situation. Survey to assess the feelings and experiences about feeding, filled by caregivers and parents.
- Well-being and withdrawal signs by the Dsilna grid : comparison during administration by parents or nurses | 6 monts
  Comparaison of the score of withdrawal or well being tube in this different situation. Survey to assess the feelings and experiences about feeding, filled by caregivers and parents.

CONTACTS AND LOCATIONS:
Overall Officials: Claire ZORES, Principal Investigator — Service de Pédiatrie, CHU de Strasbourg
Locations (1):
- Service de Pédiatrie - Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided